CLINICAL TRIAL: NCT07196670
Title: Intralesional Vitamin D Versus Intralesional Acyclovir in Plantar Warts: a Single-blinded Randomized Clinical Trial With Clinico-dermoscopic Evaluation
Brief Title: Intralesional Vitamin D Versus Intralesional Acyclovir in Plantar Warts
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Aly Abdel Aziz Gaballah, lecturer of dermatology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoUniversityKasralainy
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Plantar Warts Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): Group A will receive intralesional vitamin D3 into the base of the largest wart
  Interventions: Drug: intralesional vitamin D3 versus intralesional acyclovir
- group B (Active Comparator): Group B will receive intralesional acyclovir into the base of the largest wart
  Interventions: Drug: intralesional vitamin D3 versus intralesional acyclovir

INTERVENTIONS:
Drug: intralesional vitamin D3 versus intralesional acyclovir — injecting intralesional vitamin D in group A versus injecting intralesional acyclovir in group B in treatment of plantar warts

SUMMARY:
The goal of this clinical trial is to compare intralesional vitamin D versus intralesional acyclovir in the treatment of plantar warts. It will also learn about the safety of both techniques. The main questions it aims to answer are:

which is more effective in the treatment of plantar warts? What medical problems do participants have when taking both? What is the recurrence rate in both treatment modalities? Participants will:• Sixty plantar warts patients will be included in this study.

* They will be randomly allocated into two groups: intralesional vitamin D group (group A) and intralesional Acyclovir group (group B). Patients will be blinded to their therapeutic arm.
* All patients will be subjected to the following:

  1. Proper history taking and physical examination. Number and size of warts shall be noted.
  2. Informed consent
  3. Dermoscopic evaluation of the lesions by Fotofinder Medicam 800HD dermoscope
  4. Digital photography of the lesions
* Group A:

The aqueous solution of vitamin D3 is used (Devarol S 200,000IU/2ml ) 0.6 ml (60,000 IU ) will be slowly injected into the base of the largest wart Injections will be repeated at 3 week intervals till resolution of warts or for a maximum of 4 sessions Any hyperkeratotic lesions will be pared before injection

• Group B: Acyclovir vial (250 mg) will be diluted with 3.5 ml saline to get approximately 70 mg/ml solution 0.1 ml will be slowly injected into the base of the largest wart Injections will be repeated at 3 week intervals till resolution of warts or for a maximum of 4 sessions Any hyperkeratotic lesion will be pared before injection

• Follow up:

After cessation of treatment, there will be one month follow up during which:

* Patient will be questioned about side effects
* Physical examination to check response and/or detect recurrence
* Photography in the same positions
* Size of the warts shall be noted
* Number of warts shall be noted

  * Dermoscopic evaluation:

Patients will be examined with Fotofinder Medicam 800HD dermoscope Assessment of size and percentage of red dots and linear vessels per field At baseline, then after completion of treatment sessions and finally after 1 month from the last treatment session.

• Based on clinical, photographic and dermoscopic data, response will be graded by a blinded observer as follows: Complete response (100% disappearance of warts) Partial response (50-<100% decrease in wart size) No response (<50% decrease in wart size)

ELIGIBILITY:
Inclusion Criteria:

* patients with plantar warts, both sex, above 18 years old

Exclusion Criteria:

* under 18 years old, hypersensitivity to vitamin D or intralesional acyclovir, patients on systemic acyclovir and vitamin D, pregnant or lactating females, cognitively impaired patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
comparing the percentage of decrease in size and number of plantar warts after intralesional vitamin D versus intralesional acyclovir | 3 months

IPD SHARING:
Plan to Share IPD: Undecided